CLINICAL TRIAL: NCT04747418
Title: Uterine Inflammatory Characteristics Following Cesarean Delivery
Brief Title: Uterine Inflammatory Characteristics
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Aya Mohr-Sasson, Principal Investigator, Sheba Medical Center
Other Study IDs: 7975-20-SMC
Record Dates: First submitted 2021-01-29; First posted 2021-02-10 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Cesarean Section Complications; Fertility Disorders
Keywords: Cesarean Section Complications; Fertility Disorder; Inflammatory characteristics
MeSH Terms: interventions — Hysteroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Group: Women with low segment uterine scar following cesarean delivery: Women with low segment uterine scar following cesarean delivery, with no other abnormalities observed during diagnostic hysteroscopy
  Interventions: Procedure: Diagnostic Hysteroscopy; Procedure: Trans-vaginal ultrasound
- Cohort Group: Women with no uterine scar: Women with no uterine scar, with no other abnormalities observed during diagnostic hysteroscopy
  Interventions: Procedure: Diagnostic Hysteroscopy

INTERVENTIONS:
Procedure: Diagnostic Hysteroscopy — Collection of first 5 cc of normal saline from the output port during diagnostic hysteroscopy
Procedure: Trans-vaginal ultrasound — Trans vaginal ultrasound performed immediately following the diagnostic hysteroscopy ( as sonohysterography)
  Groups: Study Group: Women with low segment uterine scar following cesarean delivery

SUMMARY:
Data regarding fertility following niche repair is limited. It has been reported that a niche can reduce the chances of embryo implantation and may lead to spontaneous miscarriages if the implantation is close to or in the niche. One possible theory refers to inflammatory process at the area of the niche that harms the endometrial environment. Due to the aforementioned, the aim of our study is to compare the inflammatory characteristics of women with cesarean uterine scar to those without.

DETAILED DESCRIPTION:
Background As the rate of caesarean section continues to increase, concern regarding the association between delivery by caesarean section and long-term maternal morbidity has been growing . In the past decade, several articles have described a defect that can be seen on ultrasound at the site of the caesarean delivery scar, known as a 'niche' . A 'niche' describes the presence of a hypoechoic area within the myometrium of the lower uterine segment, reflecting a discontinuation of the myometrium at the site of a previous cesarean delivery. An incompletely healed scar is a long-term complication of cesarean delivery and is associated with symptoms such as postmenstrual spotting, dysmenorrhoea, chronic pelvic pain dyspareunia and subfertility. Furthermore, it can increase rates of complications during gynaecological procedures and it is associated with higher complication rate in subsequent pregnancy including: risk of rupture and morbidly adherent placenta.

Lately, a surgical resection of the abnormal myometrial area has been proposed mainly for symptomatic women, or for women that are planning future pregnancy. Different techniques have been used including hysteroscopy, laparoscopy and vaginal repair. Consideration of the surgical approach is usually determined by the patient's plans for fertility and by niche thickness. For women who do not desire pregnancy and whose niche thickness is >3 mm, a hysteroscopic approach is considered. Patients who desire future fertility, especially those with <3 mm of myometrium at the niche site, is usually recommended laparoscopic resection.

Data regarding fertility following niche repair is limited. It has been reported that a niche can reduce the chances of embryo implantation and may lead to spontaneous miscarriages if the implantation is close to or in the niche. One possible theory refers to inflammatory process at the area of the niche that harms the endometrial environment. Additional theories address the mechanical changes influencing the myometrium and the discontinuation of the endometrium at the site of the niche. Gurol Urganci et al. reported in a meta-analysis including 16 studies, that caesarean delivery reduces the probability of subsequent pregnancy by 10% [relative risk (RR) 0.91; 95% 0.87-0.95] on average, compared with a previous vaginal delivery, however, none of the studies included in the meta-analysis evaluated the relation between subsequent fertility and the presence of a niche. So far there is no definite proof for niche as a cause of infertility. Should this be supported by randomized controlled trials, it would be grounds for providing treatment that will expectedly lead to beneficial effects on reproductive outcomes. This yet needs to be proven in.

Due to the aforementioned, the aim of our study is to compare the inflammatory characteristics of women with cesarean uterine scar to those without.

Material and Methods This is a prospective study including all women visiting hysteroscopy ambulatory clinics for diagnostic hysteroscopy . All women meeting inclusion criteria will sign informed consent prior to the hysteroscopy after given explanation by one of the research team. During hysteroscopy 5 cc of the flushed water, that usually is drilled into a collecting bin that is thrown away, will be collect threw a small outlet port using a syringe connected to the outlet port of the hysteroscope. Women with normal diagnostic hysteroscopy will be included in the study. Those with low segment cesarean deliver scar will comprise the study arm and will be compared to women with no uterine scar (controls). Samples will be send to the IVF laboratory for analyzing inflammatory characteristics. Date regarding demographics, obstetrical and gynecological history will be collected from women's medical records. Primary outcome is defined as the level of inflammatory cytokines as a composite outcome

ELIGIBILITY:
Inclusion Criteria:

* Fertility age 18-45
* No abnormal finding during hysteroscopy

Exclusion Criteria:

* Women with other uterine scars (following myomectomy, T/J scar)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women with low segment uterine scar following cesarean delivery ( Study group ) and women with no uterine scar ( Controls), that have no abnormal finding on diagnostic hysterocopy.
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2025-04-07 (Actual); Study Completion 2025-04-07 (Actual)

PRIMARY OUTCOMES:
Level of inflammatory cytokines ( Granulocyte Macrophage colony stimulating factor(GM-CSF), Interferone-GAMMA, Interleukin(IL)-1,IL-2,IL-5,IL-6,IL-7,IL13,IL-15, IL-17, IL-22, IL-23,IL-31,IL-33,IL-36, Tumor Necrosis Factor (TNF) -ALPHA ) | Through study completion, an estimated period of 1 year
  All parameters will be evaluated in picogram/milliliter

SECONDARY OUTCOMES:
Niche characteristics-Residual myometrial thickness | During sonographic evaluation performed immediately following diagnostic hysteroscopy
  Evaluated in millimeters
Niche characteristics-Adjacent myometrial thickness | During sonographic evaluation performed immediately following diagnostic hysteroscopy
  Evaluated in millimeters
Niche characteristics-Depth | During sonographic evaluation performed immediately following diagnostic hysteroscopy
  Evaluated in millimeters
Niche characteristics-Length | During sonographic evaluation performed immediately following diagnostic hysteroscopy
  Evaluated in millimeters

CONTACTS AND LOCATIONS:
Overall Officials: Aya M Mohr-Sasson, M.D, Principal Investigator — Sheba Medical Center, Tel-Hashomer
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Undecided
Will be available upon request

REFERENCES:
- [Result] van der Voet LF, Bij de Vaate AM, Veersema S, Brolmann HA, Huirne JA. Long-term complications of caesarean section. The niche in the scar: a prospective cohort study on niche prevalence and its relation to abnormal uterine bleeding. BJOG. 2014 Jan;121(2):236-44. doi: 10.1111/1471-0528.12542. PMID 24373597
- [Result] Naji O, Abdallah Y, Bij De Vaate AJ, Smith A, Pexsters A, Stalder C, McIndoe A, Ghaem-Maghami S, Lees C, Brolmann HA, Huirne JA, Timmerman D, Bourne T. Standardized approach for imaging and measuring Cesarean section scars using ultrasonography. Ultrasound Obstet Gynecol. 2012 Mar;39(3):252-9. doi: 10.1002/uog.10077. PMID 21858885
- [Result] Roberge S, Boutin A, Chaillet N, Moore L, Jastrow N, Demers S, Bujold E. Systematic review of cesarean scar assessment in the nonpregnant state: imaging techniques and uterine scar defect. Am J Perinatol. 2012 Jun;29(6):465-71. doi: 10.1055/s-0032-1304829. Epub 2012 Mar 7. PMID 22399223
- [Result] Vervoort AJ, Uittenbogaard LB, Hehenkamp WJ, Brolmann HA, Mol BW, Huirne JA. Why do niches develop in Caesarean uterine scars? Hypotheses on the aetiology of niche development. Hum Reprod. 2015 Dec;30(12):2695-702. doi: 10.1093/humrep/dev240. Epub 2015 Sep 25. PMID 26409016
- [Result] Wang CB, Chiu WW, Lee CY, Sun YL, Lin YH, Tseng CJ. Cesarean scar defect: correlation between Cesarean section number, defect size, clinical symptoms and uterine position. Ultrasound Obstet Gynecol. 2009 Jul;34(1):85-9. doi: 10.1002/uog.6405. PMID 19565535
- [Result] Brown K, Tkacz Z. Hysteroscopic and laparoscopic management of caesarean scar (niche) defects in symptomatic patients. J Obstet Gynaecol. 2018 Jul;38(5):730. doi: 10.1080/01443615.2018.1444394. PMID 29944046
- [Result] Vervoort AJ, Van der Voet LF, Witmer M, Thurkow AL, Radder CM, van Kesteren PJ, Quartero HW, Kuchenbecker WK, Bongers MY, Geomini PM, de Vleeschouwer LH, van Hooff MH, van Vliet HA, Veersema S, Renes WB, van Meurs HS, Bosmans J, Oude Rengerink K, Brolmann HA, Mol BW, Huirne JA. The HysNiche trial: hysteroscopic resection of uterine caesarean scar defect (niche) in patients with abnormal bleeding, a randomised controlled trial. BMC Womens Health. 2015 Nov 12;15:103. doi: 10.1186/s12905-015-0260-8. PMID 26563197
- [Result] van der Voet LF, Vervoort AJ, Veersema S, BijdeVaate AJ, Brolmann HA, Huirne JA. Minimally invasive therapy for gynaecological symptoms related to a niche in the caesarean scar: a systematic review. BJOG. 2014 Jan;121(2):145-56. doi: 10.1111/1471-0528.12537. PMID 24373589
- [Result] Hemminki E. Impact of caesarean section on future pregnancy--a review of cohort studies. Paediatr Perinat Epidemiol. 1996 Oct;10(4):366-79. doi: 10.1111/j.1365-3016.1996.tb00062.x. PMID 8931052
- [Result] Naji O, Wynants L, Smith A, Abdallah Y, Saso S, Stalder C, Van Huffel S, Ghaem-Maghami S, Van Calster B, Timmerman D, Bourne T. Does the presence of a Caesarean section scar affect implantation site and early pregnancy outcome in women attending an early pregnancy assessment unit? Hum Reprod. 2013 Jun;28(6):1489-96. doi: 10.1093/humrep/det110. Epub 2013 Apr 12. PMID 23585560
- [Result] Gurol-Urganci I, Bou-Antoun S, Lim CP, Cromwell DA, Mahmood TA, Templeton A, van der Meulen JH. Impact of Caesarean section on subsequent fertility: a systematic review and meta-analysis. Hum Reprod. 2013 Jul;28(7):1943-52. doi: 10.1093/humrep/det130. Epub 2013 May 3. PMID 23644593
- [Result] Vissers J, Hehenkamp W, Lambalk CB, Huirne JA. Post-Caesarean section niche-related impaired fertility: hypothetical mechanisms. Hum Reprod. 2020 Jul 1;35(7):1484-1494. doi: 10.1093/humrep/deaa094. PMID 32613231
- [Result] Vitale SG, Ludwin A, Vilos GA, Torok P, Tesarik J, Vitagliano A, Lasmar RB, Chiofalo B. From hysteroscopy to laparoendoscopic surgery: what is the best surgical approach for symptomatic isthmocele? A systematic review and meta-analysis. Arch Gynecol Obstet. 2020 Jan;301(1):33-52. doi: 10.1007/s00404-020-05438-0. Epub 2020 Jan 27. PMID 31989288